CLINICAL TRIAL: NCT07402057
Title: Implementation and Evaluation of "My Care My Voice": a Program Aimed at Facilitating Conversations About Topics Such as Palliative Care
Brief Title: Implementation and Evaluation of a Program Aimed at Facilitating Palliative Care Conversations
Acronym: MCMV
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Algemeen Ziekenhuis Maria Middelares (Other); ASZ Aalst (Other); General Hospital Groeninge (Other); University Ghent (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ONZ-2025-0500; 1295225N (Other Grant/Funding Number: Research Foundation Flanders (FWO))
Record Dates: First submitted 2026-01-21; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Oncologic Diseases; Cancer
Keywords: Palliative Care; Early palliative care; Cancer; Oncology; Patient-physician communication; Patient empowerment; Health promotion; Behavioral change; Quality of life
MeSH Terms: conditions — Neoplasms; Patient Participation

STUDY DESIGN:
Intervention Model Description: Effect evaluation and process evaluation: A multicenter cluster non-equivalent controlled trial will be conducted to compare the My Care My Voice program (intervention group) with usual care (control group), including pre- and post-intervention assessments among both physicians and patients. The process evaluation will take place simultaneously with the post-intervention assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- My Care My Voice Intervention (Experimental): Participants receive the My Care My Voice intervention in addition to standard care, aimed at facilitating patient-initiated communication about palliative care between people with cancer and physicians.
  Interventions: Behavioral: My Care My Voice Intervention
- Standard care (No Intervention): Participants receive standard oncological care without the My Care My Voice intervention.

INTERVENTIONS:
Behavioral: My Care My Voice Intervention — Physicians will receive a poster, online training, and conversation card. People with cancer will receive an introductory video, poster, brochure with question and conversation cards, themed pen, and website.
  Arms: My Care My Voice Intervention

SUMMARY:
Cancer is one of the leading causes of death worldwide. In the care of people with cancer, it is essential to pay sufficient attention to individual care needs and quality of life. One component of non-cancer-directed care, care aimed at addressing symptoms independent of the cancer or tumor, may be palliative care. Palliative care can be initiated at any point along the disease trajectory and can therefore be provided simultaneously with tumor-directed care. When initiated in a timely manner, palliative care can significantly improve the quality of life of both the person living with a life-threatening condition and their family. Pain management and attention to physical, psychosocial, and spiritual needs are central to this approach. Research shows that people with cancer develop palliative care needs well before the terminal phase. Communication about care needs, and palliative care in particular, is therefore essential for the timely initiation of palliative care.

However, to date, palliative care is often initiated too late or not at all, frequently resulting in suboptimal care during the final months of life. Communication about palliative care is postponed or avoided by both healthcare professionals and people with cancer. Efforts are being made at various levels to make palliative care more discussable and to initiate it in a timely manner. At present, however, these efforts primarily focus on the role of healthcare services and professionals. By focusing solely on healthcare providers, palliative care has not yet been fully integrated as a standard component of oncological practice. The literature indicates that, in addition to barriers, there are also opportunities at the level of the person with cancer when it comes to initiating a conversation about palliative care with their physician, provided that adequate support is available.

The health promotion approach, which focuses on the role of various personal and environmental factors in stimulating healthy behavior, is well suited to addressing this need for change in patient-initiated communication about palliative care. Health promotion makes use of theoretical behavioral models, for which evidence demonstrates that their application leads to more effective behavioral interventions and successful behavior change. These models have also been shown to be promising in promoting behaviors related to palliative care and in enhancing patient empowerment.

DETAILED DESCRIPTION:
The current study aims to gain insight into the feasibility of the implementation plan of My Care My Voice (= preparation), its effectiveness in changing (the intention to) behavior (= effect evaluation), and the quality of the implementation process of the My Care My Voice intervention (= process evaluation). The study has three sub-objectives:

1. PREPARATION: A preparatory study to assess the feasibility of the implementation plan for each of the participating hospitals. Feasibility is defined as the extent to which the study is acceptable and practically feasible within the clinical setting, without imposing an excessive burden on physicians or patients. This includes:

   * The study description (aim, design, inclusion and exclusion criteria, data collection, and procedures): clarity
   * The study flow (including timeline): advantages, disadvantages, and feasibility
   * Recruitment by physicians: feasibility and support needs
   * The informed consent process: comprehensibility and clarity
   * Current workflow and consultation flow: how My Care My Voice can be integrated into existing practice → Specifically for the intervention hospitals, this includes examining how patients can be exposed to the materials (e.g., whether certain materials such as the video can be shown in the waiting room, and who - study nurse, oncology coach, etc. - can distribute materials such as the leaflet to each patient)

   In this way, facilitators can be identified, as well as potential barriers (e.g., the use of the term "palliative care" during screening and recruitment is often a reason for non-participation), allowing them to be detected and addressed in a timely manner within each specific context. This constitutes an important preparatory step toward smooth recruitment, maximal exposure to the materials, and minimal burden, all of which are key indicators of a high-quality implementation process.
2. EFFECT EVALUATION: To assess whether the My Care My Voice intervention is effective by comparing intervention hospitals with control hospitals:

   * Expected effects among physicians: Changes in behavioral determinants (intention, knowledge, attitude, self-efficacy, perceived social norm) related to responding to palliative care conversations initiated by people with cancer, and to actually engaging in these conversations with people with cancer. (The hypothesis is that My Care My Voice will positively influence these behavioral determinants, increase physicians' intention to respond to patient-initiated palliative care conversations, and lead to more actual discussions about palliative care compared with usual care.)
   * Expected effects among people with cancer: Changes in behavioral determinants (intention, knowledge, attitude, self-efficacy, perceived social norm) related to initiating a conversation about palliative care with their physician, and to actually initiating such a conversation. (The hypothesis is that My Care My Voice will positively influence these behavioral determinants, increase the intention to initiate palliative care conversations with their physician (intention = primary outcome), and result in more people with cancer actually initiating a palliative care conversation with their physician compared with usual care.)
3. PROCESS EVALUATION: To evaluate why the My Care My Voice intervention was or was not effective. The aim is to evaluate both the intervention itself and the implementation process. The process evaluation is based on the UK MRC guidelines and includes:

   * General impression: interesting, meaningful, clear
   * Implementation: extent to which instructions and guidelines were followed and adapted; what went smoothly and what did not
   * Contribution of the program: motivation, perceived impact on one's own views on palliative care (conversations) and clinical practice, perceived changes
   * Context: influence of the following factors on the course of the intervention:

Physicians: time pressure, organizational and collegial support, patient behavior, relevance of other palliative care training Patients: role/function of the person who distributed the materials, frequency of consultations, positive or negative bad news conversations

ELIGIBILITY:
Inclusion Criteria (physician):

* Oncologist (medical oncologist, radiation oncologist, etc.), radiologist, organ specialist, nuclear medicine physician, ASO
* The physician regularly interacts with people with advanced cancer
* The physician is employed in an oncology hospital department

Exclusion Criteria (physician):

* The physician works mostly (>50% of the time) in a hospital not involved in this study

Inclusion Criteria (healthcare provider - potential implementer):

* Healthcare provider (e.g., study coordinator, oncology coach) or another hospital staff member (e.g., administrative staff)
* The implementer regularly interacts with people with advanced cancer

Exclusion criteria (healthcare provider - potential implementer):

- Physician participating in My Care, My Voice

Inclusion Criteria (patient):

* The participant is an adult (18 years or older)
* The participant has been diagnosed with advanced (i.e., non-curable) cancer (no curative treatment ongoing or planned). Participants receiving life-prolonging treatment are included.
* The participant is aware of their diagnosis and treatment options as determined by their physician
* The participant has known their initial diagnosis for more than one month
* The participant is able to participate in a Dutch-language study
* The participant is competent and able to voluntarily consent to participate in this study
* The participant is hospitalized or receiving outpatient care

Exclusion Criteria (patient):

* Estimated survival prognosis by the physician is longer than 5 years
* The participant is in a follow-up trajectory or in remission according to the physician
* The participant is already receiving specialized palliative care known to the treating physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 271 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from pre-intervention measurement in the proportion of people with cancer who have a positive behavioral intention to initiate a conversation about palliative care with their physician at post-intervention measurement. | From pre-measurement to post-measurement (max. 6 months later)
  This primary outcome measure will be assessed using a study-specific self-report questionnaire developed by the research team, entitled Communication between people with cancer and their physician (Dutch language). The questionnaire will be completed by using the CAPI-method. Behavioral intention is a single item (I have the intention to start a conversation about palliative care with my physician), rated on a 5 point Likert Scale ranging from strongly disagree to strongly agree.

SECONDARY OUTCOMES:
Behavioral, psychosocial, and perceived environmental factors related to initiating a conversation about palliative care with their physician or having a positive intention to do so | From pre-measurement to post-measurement (max. 6 months later)
  These outcome measures will be assessed using a study-specific self-report questionnaire developed by the research team, entitled Communication between people with cancer and their physician (Dutch language). Behavioral factors ared measured with 120 items. The questionnaire will be completed by using the CAPI-method. Most items are rated on a 5 point Likert Scale ranging from strongly disagree to strongly agree, except of knowledge of the behavior (yes-no) and social norm (5 point Likert Scale ranging from nobody to everybody).
Behavioral, psychosocial, and perceived environmental factors related to responding to a conversation about palliative care initiated by the patient | From pre-measurement to post-measurement (12 months later)
  These outcome measures will be assessed using a study-specific self-report questionnaire developed by the research team, entitled Communication about palliative care (Dutch language). The questionnaire will be completed online. Behavioral factors are measured with 42 items. Most items are rated on a 5 point Likert Scale ranging from strongly disagree to strongly agree, except of the behavior (5 point Likert Scale ranging from never to always), knowledge about palliative care (4 point Likert Scale ranging from not correct to very correct) and social norm (5 point Likert Scale ranging from nobody to everybody).
Behavior in which people with cancer actually initiate a conversation about palliative care with their physician | From pre-measurement to post-measurement (max. 6 months later)
  This will be assessed using a study-specific self-report questionnaire developed by the research team, entitled Communication between people with cancer and their physician (Dutch language). Behavior is a single-item measure using a 5 point Likert Scale ranging from strongly disagree to strongly agree, and will also be measured based on consultation notes obtained from the electronic patient record by the treating healthcare provider.
Physicians who have a positive intention to respond to a patient-initiated conversation about palliative care | From pre-measurement to post-measurement (12 months later)
  hese outcome measures will be assessed using a study-specific self-report questionnaire developed by the research team, entitled Communication about palliative care (Dutch language). The questionnaire will be completed online. Physician behavioral intention is measured with a single item, using a 5 point Likert Scale ranging from strongly disagree to strongly agree.
Behavior in which physicians actually respond to a patient-initiated conversation about palliative care | From pre-measurement to post-measurement (12 months later)
  The behavior will be assessed using a study-specific self-report questionnaire developed by the research team, entitled Communication about palliative care (Dutch language). The questionnaire will be completed online. The physician behavior is measured with 7 items, using a 5 point Likert Scale ranging from never to always.

OTHER OUTCOMES:
Quality of life in people with incurable cancer, focusing on key symptoms and functioning using 15 questions covering physical/emotional function, pain, fatigue, appetite loss, insomnia, dyspnea, nausea/vomiting, constipation, and overall QoL | From pre-measurement to post-measurement (max. 6 months later)
  Change from pre-intervention measurement in the quality of life at the post-intervention measurement. QoL will be assessed using the EORTC QLQ-C15-PAL: 15 items using a 4 point Likert Scale ranging from not at all to very much.
Socio-demographic and medical information | From pre-measurement to post-measurement (max. 6 months later)
  These outcome measures will be assessed using both study-specific self-report questionnaire (patient + physician) developed by the research team (Dutch language).
  Patient: 9 items Physician: 13 items

CONTACTS AND LOCATIONS:
Locations (4):
- Belgium (4):
  - AZorg, Aalst, East-Flanders
  - AZ Maria Middelares, Ghent, East-Flanders
  - Ghent University Hospital, Ghent, East-Flanders
  - AZ Groeninge, Kortrijk, West-Flanders

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Scherrens AL, Cohen J, Mahieu A, Deliens L, Deforche B, Beernaert K. The perception of people with cancer of starting a conversation about palliative care: A qualitative interview study. Eur J Cancer Care (Engl). 2020 Sep;29(5):e13282. doi: 10.1111/ecc.13282. Epub 2020 Jul 1. PMID 32613675
- [Background] Scherrens AL, Beernaert K, Deliens L, Lapeire L, De Laat M, Biebuyck C, Geboes K, Van Praet C, Moors I, Deforche B, Cohen J. Identification of the most important factors related to people with cancer starting a palliative care conversation: A survey study. Psychooncology. 2022 Nov;31(11):1843-1851. doi: 10.1002/pon.6039. Epub 2022 Oct 9. PMID 36131548